CLINICAL TRIAL: NCT01265017
Title: Single-center, Double-masked, Placebo-controlled Parallel-group Study of Pregnancy-related Hormones Estradiol and Medroxyprogesterone, in Conjunction With Hydrocortisone and Growth Hormone to Stimulate C-peptide Secretion in Women With T1DM
Brief Title: Role of Pregnancy Related Hormones in Lowering the Insulin Requirement in Pregnant Women With Type 1 Diabetes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Sansum Diabetes Research Institute (Other)
Responsible Party: Principal Investigator, Kristin Castorino, DO, Principal Investigator, Sansum Diabetes Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SDRI 2009-06
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; pregnancy; insulin requirement
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Estradiol; Medroxyprogesterone; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Experimental): interventions include Estradiol, medroxyprogesterone, hydrocortisone, GH as follows
  * Estradiol 1mg every 8 hours administered orally
  * Medroxyprogesterone 2.5 mg every 24 hours administered orally
  * Hydrocortisone 2.5 mg every morning, 1.25 mg every afternoon, and 1.25 mg at bedtime administered orally
  * Growth hormone 2 mg once a day administered by subcutaneous injection
  Interventions: Drug: Estradiol, medroxyprogesterone, hydrocortisone, GH
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Estradiol, medroxyprogesterone, hydrocortisone, GH — * Estradiol 1mg every 8 hours administered orally
  * Medroxyprogesterone 2.5 mg every 24 hours administered orally
  * Hydrocortisone 2.5 mg every morning, 1.25 mg every afternoon, and 1.25 mg at bedtime administered orally
  * Growth hormone 2 mg once a day administered by subcutaneous injection,
  Other Names: estradiol,medroxyprogesterone,hydrocortisone,growth hormone
  Arms: Active Treatment
Drug: Matching placebo — matching placebo
  Other Names: inert pills
  Arms: Placebo

SUMMARY:
This is a randomized, double-masked, placebo-controlled, single-center study to evaluate stimulated C-peptide secretion after exogenous administration of mild immunosuppression and growth-promoting factors to women with preexisting T1DM who had a decline in insulin requirement or had detectable C-peptide during a previous pregnancy. Fifteen subjects will be enrolled and randomly assigned in a 2:1 ratio to either active treatment or placebo in a parallel group design.

Participation for individual subjects will consist of an initial Screening Visit, a 2-week baseline period, a Baseline Visit, visits at week 2 and 4 of the treatment period, a visit at the end of the treatment period (week 6), and a follow-up visit 2 weeks after study treatment discontinuation.

Subjects will receive either active treatment or matching placebo of estradiol 1 mg every 8 hours; medroxyprogesterone 2.5 mg every 24 hours; hydrocortisone 2.5 mg every morning, 1.25 mg every afternoon, and 1.25 mg at bedtime each night; and growth hormone 2 mg once a day).

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether women with preexisting T1DM who showed a decline in insulin requirement, defined as a decrease in insulin requirement of 25% or more, or a decrease deemed to be clinically significant by the investigator, with no other medically determined reason, or who had detectable C-peptide during a previous pregnancy will show a change in stimulated C peptide response when not pregnant and treated with exogenous pregnancy-related hormones and growth factors (Estradiol, medroxyprogesterone, hydrocortisone, GH) for 6 weeks.

The secondary objectives of this study are as follows:

* Determine whether the study treatment leads to a change in T1DM autoantibodies between Baseline and Week 6
* Determine the percentage of subjects experiencing a clinically significant decline in total daily insulin requirement at Week 6, defined as a 25% decrease from Baseline
* Descriptively evaluate the association between serum levels of growth hormone, cortisol, and prolactin and changes in C-peptide levels
* Evaluate the safety of administration of the study treatments compared with placebo, as measured by blood pressure, pulse, weight change, blood glucose, and adverse events (AEs)

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 years or older with T1DM and a documented history of at least one of the following:
* Decrease in insulin requirement with no other medically determined reason
* Detectable C-peptide
* Free of systemic corticosteroid use within 3 months before study entry.
* Stable weight (±10%)
* Stable diet and exercise
* Stable insulin requirement (<20% variability in insulin does in the 2 weeks prior to screening)Normal renal function as measured by an estimated glomerular filtration rate (simple MDRD)
* Negative pregnancy test and not planning to become pregnant during the study period. The subject must be willing to use an effective nonhormonal method of birth control during the study.
* Able to provide written informed consent.

Exclusion Criteria:

* Diagnosis of type 2 diabetes.
* Abnormal thyroid function (thyroid-stimulating hormone [TSH] and free thyroxine [FT4] test results) defined as TSH <0.4mIU/L or TSH>4.5mIU/L or Free T4 <0.6ng/dL or Free T4>1.6ng/dL.
* Abnormal renal function, as defined by serum creatinine greater than 1.2 mg/dL
* Any medical condition that, in the opinion of the investigator, yields the subject not suitable for study participation, including history of stroke, cancer, hypercoagulable problems, risk for deep vein thrombosis, and other unstable hormonal conditions, or Addison's disease or growth hormone deficiency.
* Currently treated with systemic steroids, hydrocortisone, growth hormone, or immunomodulatory medications
* Currently lactating.
* Pregnant within the last 9 months.
* Menopausal
* Taking hormonal therapy
* Known hypersensitivity to any of the medications used in this study or any component of the formulation.
* Known eating disorder
* History of phlebitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
stimulated C-peptide response | 6 weeks
  The primary efficacy endpoint is the Week 6 change from Baseline in stimulated C peptide response. It will be modeled as a function of treatment group and baseline stimulated C peptide using an analysis of covariance model. The assessment at the Screening Visit will serve as the baseline assessment in computing the C peptide change from baseline endpoint

SECONDARY OUTCOMES:
Clinical, immunologic and hormonal responses | 6 weeks
  The following secondary efficacy endpoint will be summarized descriptively and graphically by treatment group to which subjects were randomized: Week 6 changes from Baseline in the following: HbA1c, Total daily insulin requirement, IAA, GADA, IA-2A, ICA (pending the availability of sample processing, ZnT8A (pending the availability of sample processing), IGF-1, Prolactin, Growth hormone, Cortisol
Insulin requirement | 6 weeks
  Proportion of subjects with a 25% or greater decrease from Baseline in total daily insulin requirement at Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Lois Jovanovic, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States